CLINICAL TRIAL: NCT01670721
Title: A Multicenter, Single Arm, Open Label Clinical Trial Evaluating Safety and Health Related Quality of Life of Aflibercept in Combination With Irinotecan/5-FU Chemotherapy (FOLFIRI) in Patients With Metastatic Colorectal Cancer (mCRC) Previously Treated With an Oxaliplatin-Containing Regimen
Brief Title: Colorectal Cancer Metastatic
Acronym: AFEQT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFLIBL06266; 2012-000048-89; U1111-1128-9325 (Other: UTN)
Record Dates: First submitted 2012-07-13; First posted 2012-08-22 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — aflibercept; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin) (Experimental): Aflibercept 4 mg/kg intravenous (IV) infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until DP, unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
  Interventions: Drug: AFLIBERCEPT; Drug: Irinotecan; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: AFLIBERCEPT — Pharmaceutical form:Concentrate for solution for infusion; Route of administration: Intravenous
  Other Names: AVE0005
Drug: Irinotecan — Pharmaceutical form:Concentrate for solution for infusion; Route of administration: Intravenous
Drug: Fluorouracil — Pharmaceutical form:Concentrate for solution for infusion; Route of administration: Intravenous
Drug: Leucovorin — Pharmaceutical form:Concentrate for solution for infusion; Route of administration: Intravenous

SUMMARY:
Primary Objective:

To evaluate the safety of aflibercept in participants with mCRC treated with irinotecan/5-Fluorouracil (5-FU) combination (FOLFIRI) after failure of an oxaliplatin-based regimen (participants similar to those evaluated in the VELOUR trial [EFC10262, NCT00561470]) according to side effects prevention and management guidelines.

Secondary Objective:

To document the Health-Related Quality of Life (HRQL) of aflibercept in this participant population.

DETAILED DESCRIPTION:
Each participant was treated until disease progression (DP), unacceptable toxicity, death, Investigator's decision or participant's refusal for further treatment (whichever come first). Participants were followed-up during treatment and for at least 30 days after its last study treatment (either Aflibercept or FOLFIRI) administration, up to a maximum of 6 months.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum.
* Metastatic disease.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* One and only one prior chemotherapeutic regimen for metastatic disease. This prior chemotherapy must be an oxaliplatin containing regimen. Participants must progressed during or following the last administration of the oxaliplatin based chemotherapy. Participants relapsing within 6 months of completion of oxaliplatin adjuvant chemotherapy were also eligible.
* Participants must be affiliated to a Social Security System.

Exclusion criteria:

Related to Methodology

* Prior therapy with irinotecan; Absolute neutrophil counts (ANC) <1.5 x 109/L; Platelet count <100 x 109/L; Hemoglobin <9.0 g/dL; Total bilirubin >1.5 x upper limit of normal (ULN); Transaminases >3 x ULN (unless liver metastasis are present, 5 x ULN in that case); Alkaline phosphatase >3 x ULN (unless liver metastasis are present, 5 x ULN in that case).
* Less than 4 weeks elapsed from prior radiotherapy or prior chemotherapy or major surgery to the time of inclusion or until the surgical wound was fully healed whichever came later (48 hours in case of minor surgical procedure or until wound full healing observed).
* Treatment with any investigational drug within 30 days prior to inclusion.
* AEs (with exception of alopecia, peripheral sensory neuropathy and those listed in specific exclusion criteria) from any prior anti cancer therapy of grade >1 National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v.4.0 at the time of inclusion.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Other prior malignancy. Basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or any other cancer from which the participant had been disease free for >5 years were allowed.
* Any of the following within 6 months prior to inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior to inclusion: Grade 3-4 gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event.
* Occurrence of deep vein thrombosis within 4 weeks, prior to inclusion.
* Known acquired immunodeficiency syndrome (AIDS)-related illnesses or known human deficiency virus (HIV) disease requiring antiretroviral treatment.
* Any severe acute or chronic medical condition, which could impair the ability of the participant to participate to the study or to interfere with interpretation of study results.
* Pregnant or breast-feeding women. Positive pregnancy test for women of reproductive potential.
* Participants with reproductive potential (female and male) who did not agree to use a method of contraception during the study treatment period and for at least 6 months following completion of study treatment. The definition of effective method was left to the investigator's judgment.

Related to Aflibercept:

* Urine protein-creatinine ratio (UPCR) >1 on morning spot urinalysis or proteinuria > 500 mg/24-h.
* Serum creatinine >1.5 x ULN . If creatinine 1.0-1.5 x ULN, creatinine clearance, calculated according to Cockroft-Gault formula, <60 ml/min will exclude the participant.
* Uncontrolled hypertension (blood pressure >140/90 mmHg or systolic blood pressure >160 mmHg when diastolic blood pressure <90 mmHg, on at least 2 repeated determinations on separate days, or upon clinical judgement within 3 months prior to study inclusion.
* Participants on anticoagulant therapy with unstable dose of warfarin and/or having an out-of-therapeutic range international normalized ratio (INR) (>3) within the 4 weeks prior to inclusion.
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy (e.g. INR >1.5 without vitamine K antagonist therapy), non-healing wound.

Related to FOLFIRI

* Known dihydropyrimidine dehydrogenase deficiency.
* Predisposing colonic or small bowel disorders in which the symptoms were uncontrolled as indicated by baseline of >3 loose stools daily.
* Prior history of chronic enteropathy, inflammatory enteropathy, chronic diarrhea, unresolved bowel obstruction/sub-obstruction, more than hemicolectomy, extensive small intestine resection with chronic diarrhea.
* History of anaphylaxis or known intolerance to atropine sulphate or loperamide or appropriate antiemetics to be administered in conjunction with FOLFIRI.
* Treatment with concomitant anticonvulsivant agents that are cytochrome P450 3A4 (CYP3A4) inducers (phenytoin, phenobarbital, carbamazepine), unless discontinued >7 days.
* Participants with known Gilbert's syndrome.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative office, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 38 sites in France. A total of 182 participants were screened between 08 August 2012 and 30 June 2014, out of which 175 participants were enrolled and treated.
Pre-assignment Details: Participants enrolled in the study to assess the safety of Aflibercept in participants treated with a combination of Aflibercept with FOLFIRI regimen (Irinotecan, Leucovorin and 5-Fluorouracil [5-FU]).
Groups:
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin): Aflibercept 4 mg/kg intravenous (IV) infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until disease progression (DP), unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
Period: Overall Study
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Started | 175
Completed | 122 (81 participants with DP and 41 with adverse events were considered as completed.)
Not Completed | 53
Not completed — Participant's decision | 15
Not completed — Other than specified above | 38

BASELINE CHARACTERISTICS:
Groups:
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin): Aflibercept 4 mg/kg IV infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until DP, unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period. On-treatment period was defined as the time from the first dose of treatment to 30 days after the last dose of treatment (either Aflibercept or FOLFIRI). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline upto 30 days after the last treatment administration (either Aflibercept or FOLFIRI whichever comes last) (maximum exposure:723 days)
Population: Safety population defined as the participants who signed the informed consent form and received at least part of one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 175
Percentage of participants
  Any TEAE | 100.00
  Any serious TEAE | 40.6
  Any serious related TEAE | 21.1
  Any TEAE leading to death | 9.1
  Any TEAE (permanent treatment discontinuation) | 23.4
  Any TEAE (premature treatment discontinuation) | 16.0

2. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) European Organization for Research and Treatment for Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) & other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favorable outcome with a best quality of life for participant.
Time Frame: Pre-dose at Baseline, Day 1 of every odd cycle; and at end of treatment (30 days after last study treatment) (maximum exposure: 99 weeks)
Population: EORTC QLQ-C30 analysis population: participants who signed informed consent form; had an evaluable QLQ-C30 questionnaire at baseline and at least one evaluable assessment post baseline and received at least part of one dose of study treatment(either Aflibercept or FOLFIRI).Here, n=number of participants with available data at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 152
units on a scale
  Baseline (n=148) | 69.54 (18.97)
  At Cycle 3 (n=130) | -7.56 (19.78)
  At Cycle 5 (n=99) | -10.86 (19.76)
  At Cycle 7 (n=72) | -8.22 (20.00)
  At Cycle 9 (n=51) | -9.31 (19.34)
  At Cycle 11 (n=45) | -14.81 (21.24)
  At Cycle 13 (n=25) | -12.67 (24.31)
  At Cycle 15 (n=24) | -12.50 (18.22)
  At Cycle 17 (n=14) | -14.29 (15.82)
  At Cycle 19 (n=12) | -15.28 (11.70)
  At Cycle 21 (n=10) | -15.83 (19.82)
  At Cycle 23 (n=6) | -9.72 (20.01)
  At Cycle 25 (n=4) | -8.33 (6.80)
  At Cycle 27 (n=4) | -12.50 (15.96)
  At Cycle 29 (n=2) | -8.33 (11.79)
  At Cycle 31 (n=2) | -16.67 (0.00)
  At Cycle 33 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 33, standard deviation could not be calculated.
  At Cycle 35 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 35, standard deviation could not be calculated.
  At Cycle 37 (n=2) | -8.33 (11.79)
  At Cycle 39 (n=2) | -8.33 (11.79)
  At Cycle 41 (n=2) | -8.33 (11.79)
  At Cycle 43 (n=2) | -12.50 (5.89)
  At Cycle 45 (n=2) | -4.17 (17.68)
  At Cycle 47 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 47, standard deviation could not be calculated.
  At end of study treatment (n=73) | -11.19 (24.38)

3. Secondary Outcome: Change From Baseline in HRQL European-Quality of Life-5 Dimension Instrument-3 Levels (EQ-5D-3L) Index Score
Description: EQ-5D was a standardized HRQL questionnaire consisting of EQ-5D descriptive system and Visual Analogue Scale (VAS). EQ-5D descriptive system comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on 3 levels (no problem, some problems & severe problems) within a particular EQ-5D dimension. 5 dimensional 3-level system was converted into single index utility score. Possible values for single index utility score ranged from -0.594 (severe problems in all dimensions) to 1.0 (no problem in all dimensions) on scale where 1 represented best possible health state.
Time Frame: as for outcome 2
Population: EQ-5D analysis population: participants who signed informed consent form, had an evaluable EQ-5D questionnaire at baseline and at least one evaluable assessment post baseline and received at least part of one dose of study treatment (either Aflibercept or FOLFIRI).Here, n = number of participants with available data at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 148
units on a scale
  Baseline (n=148) | 0.78 (0.21)
  At Cycle 3 (n=127) | -0.04 (0.23)
  At Cycle 5 (n=96) | -0.08 (0.25)
  At Cycle 7 (n=72) | -0.05 (0.20)
  At Cycle 9 (n=49) | -0.09 (0.23)
  At Cycle 11 (n=43) | -0.06 (0.20)
  At Cycle 13 (n=24) | -0.09 (0.14)
  At Cycle 15 (n=25) | -0.10 (0.16)
  At Cycle 17 (n=14) | -0.03 (0.10)
  At Cycle 19 (n=12) | -0.10 (0.12)
  At Cycle 21 (n=10) | -0.03 (0.18)
  At Cycle 23 (n=6) | -0.08 (0.15)
  At Cycle 25 (n=3) | 0.04 (0.22)
  At Cycle 27 (n=3) | -0.09 (0.20)
  At Cycle 29 (n=2) | -0.18 (0.04)
  At Cycle 31 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 31, standard deviation could not be calculated.
  At Cycle 37 (n=1) | -0.15 (NA) — As only one participant was analyzed at cycle 37, standard deviation could not be calculated.
  At Cycle 39 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 39, standard deviation could not be calculated.
  At Cycle 41 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 41, standard deviation could not be calculated.
  At Cycle 43 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 43, standard deviation could not be calculated.
  At Cycle 45 (n=1) | 0.00 (NA) — As only one participant was analyzed at cycle 45, standard deviation could not be calculated.
  At end of study treatment (n=71) | -0.20 (0.31)

4. Secondary Outcome: Change From Baseline in HRQL EQ-5D-3L VAS Score
Description: EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state. Baseline corresponded to last evaluable assessment before treatment administration.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 148
units on a scale
  Baseline (n=125) | 69.48 (19.10)
  At cycle 3 (n=94) | -6.23 (17.82)
  At cycle 5 (n=76) | -7.62 (17.23)
  At cycle 7 (n=57) | -7.79 (14.14)
  At cycle 9 (n=38) | -7.55 (16.12)
  At cycle 11 (n=36) | -8.67 (16.09)
  At cycle 13 (n=22) | -8.95 (17.56)
  At cycle 15 (n=22) | -12.41 (19.57)
  At cycle 17 (n=13) | -10.31 (17.44)
  At cycle 19 (n=10) | -15.70 (18.19)
  At cycle 21 (n=8) | -15.13 (19.87)
  At cycle 23 (n=5) | -8.80 (10.71)
  At cycle 25 (n=2) | -13.00 (4.24)
  At cycle 27 (n=3) | -15.67 (9.81)
  At cycle 29 (n=2) | -17.50 (3.54)
  At cycle 31 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 31, standard deviation could not be calculated.
  At cycle 37 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 37, standard deviation could not be calculated.
  At cycle 39 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 39, standard deviation could not be calculated.
  At cycle 41 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 41, standard deviation could not be calculated.
  At cycle 43 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 43, standard deviation could not be calculated.
  At cycle 45 (n=1) | -15.00 (NA) — As only one participant was analyzed at cycle 45, standard deviation could not be calculated.
  At end of study treatment (n=55) | -13.05 (20.82)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 723) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment-emergent that is AEs that developed/worsened and deaths that occurred during 'on-treatment period' (from the first dose of treatment to 30 days after the last dose of treatment [either aflibercept or FOLFIRI]).
Groups:
- Aflibercept + FOLFIRI(Irinotecan, 5-Fluorouracil & Leucovorin): Aflibercept 4 mg/kg IV infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until DP, unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment (maximum exposure: Week 99).
Arm/Group | Aflibercept + FOLFIRI(Irinotecan, 5-Fluorouracil & Leucovorin)
Serious Adverse Events (participants affected / at risk) | 71/175
Other Adverse Events (participants affected / at risk) | 172/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI(Irinotecan, 5-Fluorouracil & Leucovorin) (N=175)
ANAEMIA (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
VITREOUS HAEMORRHAGE (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ANAL FISTULA (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 8
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 2
PANCREATITIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
RECTOURETHRAL FISTULA (Gastrointestinal disorders) | 1
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 2
TOOTH LOSS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
DISEASE PROGRESSION (General disorders) | 9
FATIGUE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 8
INFLUENZA LIKE ILLNESS (General disorders) | 1
PYREXIA (General disorders) | 3
HEPATIC FAILURE (Hepatobiliary disorders) | 2
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
DEVICE RELATED SEPSIS (Infections and infestations) | 1
ESCHERICHIA INFECTION (Infections and infestations) | 1
INFECTION (Infections and infestations) | 2
LUNG INFECTION (Infections and infestations) | 2
PELVIC ABSCESS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1
LAPAROSCOPY (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBELLAR ISCHAEMIA (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
URINARY RETENTION (Renal and urinary disorders) | 1
PRIAPISM (Reproductive system and breast disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
HEPATECTOMY (Surgical and medical procedures) | 1
INTRAPERITONEAL HYPERTHERMIC CHEMOTHERAPY (Surgical and medical procedures) | 1
PHLEBITIS (Vascular disorders) | 1
THROMBOSIS (Vascular disorders) | 1
VARICOSE ULCERATION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI(Irinotecan, 5-Fluorouracil & Leucovorin) (N=175)
NEUTROPENIA (Blood and lymphatic system disorders) | 39
ABDOMINAL PAIN (Gastrointestinal disorders) | 36
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 14
CONSTIPATION (Gastrointestinal disorders) | 39
DIARRHOEA (Gastrointestinal disorders) | 121
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 10
NAUSEA (Gastrointestinal disorders) | 86
PROCTALGIA (Gastrointestinal disorders) | 10
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 11
STOMATITIS (Gastrointestinal disorders) | 83
VOMITING (Gastrointestinal disorders) | 47
ASTHENIA (General disorders) | 98
FATIGUE (General disorders) | 33
PYREXIA (General disorders) | 14
WEIGHT DECREASED (Investigations) | 68
DECREASED APPETITE (Metabolism and nutrition disorders) | 59
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18
MYALGIA (Musculoskeletal and connective tissue disorders) | 11
DYSGEUSIA (Nervous system disorders) | 13
HEADACHE (Nervous system disorders) | 32
NEUROPATHY PERIPHERAL (Nervous system disorders) | 19
PARAESTHESIA (Nervous system disorders) | 9
PROTEINURIA (Renal and urinary disorders) | 25
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 22
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 43
ALOPECIA (Skin and subcutaneous tissue disorders) | 36
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 23
HYPERTENSION (Vascular disorders) | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.